CLINICAL TRIAL: NCT05374369
Title: Retrospective Analysis of Colorectal Cancer Screening Results Among People Aged 40-74 in Shipai Town, Dongguan City, China
Brief Title: Retrospective Analysis of Colorectal Cancer Screening Results
Status: Completed | Type: Observational
Sponsor: Creative Biosciences (Guangzhou) Co., Ltd. (Industry)
Collaborators: Dongguan Shipai Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: KLM2021-03
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer; Advanced Adenocarcinoma; Hyperplastic Polyp; Colorectal Neoplasms; Digestive System Neoplasm; Neoplasms
Keywords: Colorectal Cancer; Colon Cancer; Stool DNA test; Fecal DNA test; Fecal Immunochemical Test; FIT; Methylation Biomarkers; Colonoscopy; Cancer Screening
MeSH Terms: conditions — Colorectal Neoplasms; Digestive System Neoplasms; Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subjects with positive SDC2 Gene Methylation Test: Subjects must meet both of the following criteria to be eligible for the study:
  1. Subjects with positive SDC2 Gene Methylation Test;
  2. Subjects with colonoscopy results and/or pathological results.
  Interventions: Diagnostic Test: SDC2 Gene Methylation Test and Q-FIT Test; Procedure: Colonoscopy and/or pathological examination
- Subjects with positive Q-FIT Test: Subjects must meet both of the following criteria to be eligible for the study:
  1. Subjects with positive Q-FIT Test;
  2. Subjects with colonoscopy results and/or pathological results.
  Interventions: Diagnostic Test: SDC2 Gene Methylation Test and Q-FIT Test; Procedure: Colonoscopy and/or pathological examination
- Subjects with positive SDC2 Gene Methylation Test and Q-FIT Test: Subjects must meet both of the following criteria to be eligible for the study:
  1. Subjects with positive SDC2 Gene Methylation Test and Q-FIT Test;
  2. Subjects with colonoscopy results and/or pathological results.
  Interventions: Diagnostic Test: SDC2 Gene Methylation Test and Q-FIT Test; Procedure: Colonoscopy and/or pathological examination

INTERVENTIONS:
Diagnostic Test: SDC2 Gene Methylation Test and Q-FIT Test — Stool specimens were collected by the subjects for SDC2 Gene Methylation Test and Q-FIT Test
Procedure: Colonoscopy and/or pathological examination — Subjects underwent colonoscopy and/or pathological examination.

SUMMARY:
The purpose of this study is to retrospectively analyze colorectal cancer screening data of 40-74 year old population in Shipai Town, Dongguan City.

In this study, the data of SDC2 Gene Methylation Test and Fecal Immunochemistry Test (Q-FIT) were screened from about 11,000 subjects who participated in Colorectal Cancer Screening in Shipai Town People's Livelihood Project from May 2021 to May 2022. Data from 822 subjects with positive SDC2 Gene Methylation Test and/or positive Fecal Immunochemistry Test (Q-FIT) results and with colonoscopy and/or pathological results were selected for retrospective analysis.

This retrospective study evaluated the screening performance of SDC2 Gene Methylation Test and/or Fecal Immunochemistry Test (Q-FIT) for colorectal cancer using colonoscopy and/or pathological results as the clinical standard method.

DETAILED DESCRIPTION:
This study is a retrospective and observational study. Subjects were not be given or offered any treatment during the study. The investigator reviewed the patient's medical history and examination report to determine eligibility based on inclusion and exclusion criteria.

This study retrospectively analyse the basic information and the test results of SDC2 Gene Methylation Test and Fecal Immunochemistry Test (Q-FIT) of about 11,000 subjects who participated in the Colorectal Cancer Screening in Shipai Town People's Livelihood Project from May 2021 to May 2022. A total of 822 subjects with positive SDC2 Gene Methylation Test results and / or positive Fecal Immunochemistry Test (Q-FIT) results were screened out and their colonoscopy results were collected.

822 subjects were classified according to colonoscopy and/or pathological detection results, and the screening performance of the SDC2 Gene Methylation Test and Fecal Immunochemistry Test (Q-FIT) for colorectal cancer was statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet both of the following criteria to be eligible for the study:

1. Subjects with positive SDC2 Gene Methylation Test and/or Q-FIT;
2. Subjects with colonoscopy and/or pathological results.

Exclusion Criteria:

Subject with any of the following conditions shall be excluded:

1. Data Missing or damaged;
2. Unqualified colonoscopy or unqualified stool test.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects live in Shipai Town, Dongguan city, the age limit is 40-74 years，822 subjects meet the inclusion criteria for this study.
Sampling Method: Non-Probability Sample
Enrollment: 822 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Positive predictive value (PPV) | one month
  PPV is the number of real positive cases in the total number of stool gene DNA methylation detection positive or/and Q-FIT positive.
Sensitivity | one month
  Sensitivity is the percentage of subjects with colon cancer who are correctly identified by the testing kit.
Tumor detection rate in the positive screening results | one month
  Compare to clinical standard method results, the tumor detection rates of the three groups were analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi Zhang, Principal Investigator — Dongguan Shipai Hospital
Locations (1):
- Dongguan Shipai Hospital, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
We are carefully considering all applicable regulations and laws governing sharing of patients' data from China online with the global public.

REFERENCES:
- [Derived] Kong X, Wu Q, Zhang Z, Yu Z, Niu F, Wang X, Zou H. Effectiveness of single-target fecal DNA methylation test in regional mass screening for colorectal cancer and precancerous lesions in China. Gastroenterol Rep (Oxf). 2025 Apr 15;13:goaf029. doi: 10.1093/gastro/goaf029. eCollection 2025. PMID 40241850